CLINICAL TRIAL: NCT01665144
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Variable Treatment Duration Study Evaluating the Efficacy and Safety of Siponimod (BAF312) in Patients With Secondary Progressive Multiple Sclerosis Followed by Extended Treatment With Open-label BAF312.
Brief Title: Exploring the Efficacy and Safety of Siponimod in Patients With Secondary Progressive Multiple Sclerosis (EXPAND)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBAF312A2304; 2012-003056-36 (EudraCT Number)
Record Dates: First submitted 2012-08-03; First posted 2012-08-15 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — siponimod

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Siponimod (BAF312) (Experimental): Participants started on Day 1 and were uptitrated from 0.25 mg to 2 mg of BAF312 orally over a period of 6 days. After Day 7, participants continued on the treatment epoch for 3 months. During the Core Part of the study, participants participated in a maximum of 3 epochs. Following the Core Part, eligible patients enter the Extension Part during which all receive open-label BAF312.
  Interventions: Drug: BAF312
- Placebo (Placebo Comparator): Matching placebo to BAF312 was administered orally during the Core Part of the trial. Following the Core Part, eligible participants enter the Extension Part during which all receive open-label BAF312.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAF312 — 0.25, 0.5, 1, and 2 mg film-coated tablets
  Arms: Siponimod (BAF312)
Drug: Placebo — Film-coated tablets
  Arms: Placebo

SUMMARY:
Evaluate the safety and efficacy of Siponimod (BAF312) versus placebo in a variable treatment duration in patients with secondary progressive multiple sclerosis (Core Part) followed by extended treatment with open-label BAF312 to obtain data on long-term safety, tolerability and efficacy (Extension Part).

DETAILED DESCRIPTION:
This study had two parts, a Core Part and an Extension Part. The Core Part of the study was a randomized, multicenter, double-blind, placebo-controlled parallel-group study in patients with secondary progressive multiple sclerosis (SPMS). Eligible patients were randomized (2:1) to receive either siponimod or placebo. The duration of the Core Part of the study was variable for each patient, given that this was an event-driven study and terminated when a pre-defined number of confirmed disability progression (CDP) events had occurred irrespective of duration of individual patient participation. Patients who had 6-month CDP during the Treatment Epoch of the Core Part were provided with options that included starting treatment with open label siponimod as rescue medication.

Patients who were eligible to enter the Extension Part received open label siponimod.

ELIGIBILITY:
Inclusion Criteria:

* Prior history of relapsing remitting MS
* SPMS defined as progressive increase of disability over at least 6 months
* EDSS score of 3.0 to 6.5
* No relapse of corticosteroid treatment within 3 months

Exclusion Criteria:

* Women of child bearing potential must use reliable forms of contraception.
* Diagnosis of Macular edema during screening period
* Any medically unstable condition determined by investigator.
* Unable to undergo MRI scans
* Hypersensitivity to any study drugs or drugs of similar class

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1651 (Actual)
Dates: Start 2012-12-20 (Actual); Primary Completion 2016-04-29 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (252):
- United States (48):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Berkeley, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Basalt, Colorado
  - Novartis Investigative Site, Boulder, Colorado
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Englewood, Colorado
  - Novartis Investigative Site, Fairfield, Connecticut
  - Novartis Investigative Site, Delray Beach, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Maitland, Florida
  - Novartis Investigative Site, Ormond Beach, Florida
  - Novartis Investigative Site, Port Charlotte, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Vero Beach, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Evanston, Illinois
  - Novartis Investigative Site, Flossmoor, Illinois
  - Novartis Investigative Site, Lenexa, Kansas
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Plymouth, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, Freehold, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Patchogue, New York
  - Novartis Investigative Site, Stony Brook, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Springfield, Oregon
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Lubbock, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Burlington, Vermont
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
- Australia (5):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Austria (2):
  - Novartis Investigative Site, Klagenfurt
  - Novartis Investigative Site, Vienna
- Belgium (8):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Fraiture En Condroz, Belgium
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Overpelt
  - Novartis Investigative Site, Sijsele
- Bulgaria (2):
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (9):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Burnaby, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
- China (6):
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Czechia (4):
  - Novartis Investigative Site, Brno, Czech Rep.
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Jihlava
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Tallinn, Estonia
- France (11):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nancy
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Strasbourg
- Germany (40):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Bad Mergentheim
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Itzehoe
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neuburg an der Donau
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Prien am Chiemsee
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Schwendi
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Stadtroda
  - Novartis Investigative Site, Teupitz
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Unterhaching
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Würzburg
- Greece (3):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Heraklion Crete
  - Novartis Investigative Site, Thessaloniki
- Hungary (8):
  - Novartis Investigative Site, Budapest, HUN
  - Novartis Investigative Site, Esztergom, HUN
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Veszprém
- Novartis Investigative Site, Dublin, Ireland
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Italy (5):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Cefalù, PA
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Japan (14):
  - Novartis Investigative Site, Tōon, Ehime
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Morioka, Iwate
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Kawagoe, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Aomori
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Osaka
- Latvia (2):
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Riga
- Lithuania (3):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Vilnius
- Netherlands (6):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Hoorn
  - Novartis Investigative Site, Sittard-Geleen
  - Novartis Investigative Site, Tilburg
- Poland (8):
  - Novartis Investigative Site, Gmina Końskie
  - Novartis Investigative Site, Grudziądz
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Portugal (5):
  - Novartis Investigative Site, Amadora
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Romania (5):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Constanța
  - Novartis Investigative Site, Suceava
  - Novartis Investigative Site, Târgu Mureş
  - Novartis Investigative Site, Timișoara
- Russia (6):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Ufa
- Slovakia (7):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Martin
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Trenčín
  - Novartis Investigative Site, Trnava
- Spain (12):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
- Switzerland (7):
  - Novartis Investigative Site, Aarau, CH
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Lucerne
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Zurich
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Altunizade
  - Novartis Investigative Site, Haseki Istanbul
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Mecidiyekoy Istanbul
  - Novartis Investigative Site, Samsun
  - Novartis Investigative Site, Trabzon
- United Kingdom (9):
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Headington, Oxfordshire
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
  Locations: central Contact Info Novartis.email@novartis.com

REFERENCES:
- [Derived] Gold R, Piani-Meier D, Kappos L, Bar-Or A, Vermersch P, Giovannoni G, Fox RJ, Arnold DL, Benedict RHB, Penner IK, Rouyrre N, Kilaru A, Karlsson G, Ritter S, Dahlke F, Hach T, Cree BAC. Siponimod vs placebo in active secondary progressive multiple sclerosis: a post hoc analysis from the phase 3 EXPAND study. J Neurol. 2022 Sep;269(9):5093-5104. doi: 10.1007/s00415-022-11166-z. Epub 2022 May 31. PMID 35639197
- [Derived] Cree BA, Arnold DL, Fox RJ, Gold R, Vermersch P, Benedict RH, Bar-Or A, Piani-Meier D, Rouyrre N, Ritter S, Kilaru A, Karlsson G, Giovannoni G, Kappos L. Long-term efficacy and safety of siponimod in patients with secondary progressive multiple sclerosis: Analysis of EXPAND core and extension data up to >5 years. Mult Scler. 2022 Sep;28(10):1591-1605. doi: 10.1177/13524585221083194. Epub 2022 Apr 5. PMID 35380078
- [Derived] Leppert D, Kropshofer H, Haring DA, Dahlke F, Patil A, Meinert R, Tomic D, Kappos L, Kuhle J. Blood Neurofilament Light in Progressive Multiple Sclerosis: Post Hoc Analysis of 2 Randomized Controlled Trials. Neurology. 2022 May 24;98(21):e2120-e2131. doi: 10.1212/WNL.0000000000200258. Epub 2022 Apr 4. PMID 35379762
- [Derived] Arnold DL, Piani-Meier D, Bar-Or A, Benedict RH, Cree BA, Giovannoni G, Gold R, Vermersch P, Arnould S, Dahlke F, Hach T, Ritter S, Karlsson G, Kappos L, Fox RJ; EXPAND Clinical Investigators. Effect of siponimod on magnetic resonance imaging measures of neurodegeneration and myelination in secondary progressive multiple sclerosis: Gray matter atrophy and magnetization transfer ratio analyses from the EXPAND phase 3 trial. Mult Scler. 2022 Sep;28(10):1526-1540. doi: 10.1177/13524585221076717. Epub 2022 Mar 9. PMID 35261318
- [Derived] Schur N, Gudala K, Vudumula U, Vadapalle S, Bhadhuri A, Casanova A, Adlard N, Schwenkglenks M. Cost Effectiveness and Budget Impact of Siponimod Compared to Interferon Beta-1a in the Treatment of Adult Patients with Secondary Progressive Multiple Sclerosis with Active Disease in Switzerland. Pharmacoeconomics. 2021 May;39(5):563-577. doi: 10.1007/s40273-021-01023-8. Epub 2021 Apr 1. PMID 33791945
- [Derived] Benedict RHB, Tomic D, Cree BA, Fox R, Giovannoni G, Bar-Or A, Gold R, Vermersch P, Pohlmann H, Wright I, Karlsson G, Dahlke F, Wolf C, Kappos L. Siponimod and Cognition in Secondary Progressive Multiple Sclerosis: EXPAND Secondary Analyses. Neurology. 2021 Jan 19;96(3):e376-e386. doi: 10.1212/WNL.0000000000011275. Epub 2020 Dec 16. PMID 33328324
- [Derived] Kappos L, Bar-Or A, Cree BAC, Fox RJ, Giovannoni G, Gold R, Vermersch P, Arnold DL, Arnould S, Scherz T, Wolf C, Wallstrom E, Dahlke F; EXPAND Clinical Investigators. Siponimod versus placebo in secondary progressive multiple sclerosis (EXPAND): a double-blind, randomised, phase 3 study. Lancet. 2018 Mar 31;391(10127):1263-1273. doi: 10.1016/S0140-6736(18)30475-6. Epub 2018 Mar 23. PMID 29576505

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 294 investigative sites in 31 countries.
Pre-assignment Details: Core Part recruitment completed; eligible patients moved to Extension Part (EP) providing treatment up to additional 7 years. Projected full 7-year final visits for majority patients first quarter 2023. Novartis closed EP slightly earlier than planned (not based on safety issues) to accommodate changes in study operations at a point when objective to provide long-term safety/efficacy data in patients treated up to 7 years met. Consequently, EP considered completed.
Groups:
- Siponimod (BAF312): Participants started on Day 1 and were uptitrated from 0.25 mg to 2 mg of BAF312 orally over a period of 6 days. After Day 7, participants continued on 2 mg BAF312 daily for a variable duration.
- Placebo: Matching placebo to BAF312 was administered orally during the Core Part of the trial.
- Placebo-BAF312: Participants who received placebo in the Core Part and switched to siponimod in the Extension Part.
Period: Core Part
Arm/Group | Siponimod (BAF312) | Placebo | Placebo-BAF312
Started (All randomized patients.) | 1105 | 546 | 0
Safety Set (All patients who received at least one dose of study medication. Patients were analyzed according to the actual treatment received.) | 1099 | 546 | 0
Full Analysis Set (All randomized patients with assigned treatments who took at least one dose of study medication. Patients were analyzed according to the randomized treatment assignment.) | 1099 | 546 | 0
Completed | 903 | 424 | 0
Not Completed | 202 | 122 | 0
Not completed — Withdrawal by Subject | 96 | 77 | 0
Not completed — Adverse Event | 45 | 18 | 0
Not completed — Lack of Efficacy | 16 | 11 | 0
Not completed — Lost to Follow-up | 9 | 8 | 0
Not completed — Physician Decision | 13 | 1 | 0
Not completed — Progressive disease | 8 | 4 | 0
Not completed — Non-compliance with study treatment | 5 | 0 | 0
Not completed — Death | 3 | 1 | 0
Not completed — Protocol deviation | 3 | 1 | 0
Not completed — New therapy for study indication | 2 | 1 | 0
Not completed — Technical problems | 2 | 0 | 0
Period: Extension Part
Arm/Group | Siponimod (BAF312) | Placebo | Placebo-BAF312
Started | 821 | 0 | 399
Completed | 326 | 0 | 159
Not Completed | 495 | 0 | 240
Not completed — Patient/guardian decision | 180 | 0 | 98
Not completed — Adverse Event | 104 | 0 | 59
Not completed — Study closed early | 42 | 0 | 19
Not completed — Progressive disease | 36 | 0 | 14
Not completed — Lack of Efficacy | 37 | 0 | 12
Not completed — Physician Decision | 29 | 0 | 13
Not completed — Technical problems | 20 | 0 | 8
Not completed — Death | 20 | 0 | 4
Not completed — Missing | 12 | 0 | 6
Not completed — Lost to Follow-up | 9 | 0 | 5
Not completed — New therapy for study indication | 3 | 0 | 2
Not completed — Protocol deviation | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Siponimod (BAF312) | Placebo | Total
Number analyzed (Participants) | 1105 | 546 | 1651
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.0 (7.84) | 48.1 (7.94) | 48.0 (7.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 669 | 323 | 992
  Male | 436 | 223 | 659
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 31 | 18 | 49
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 1050 | 513 | 1563
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 3-month Confirmed Disability Progression (CDP) Events as Measured by the Expanded Disability Status Scale (EDSS)
Description: The EDSS uses an ordinal scale to assess neurologic impairment in MS based on a neurological examination. Scores in each of 7 functional systems (Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel & Bladder, and Cerebral) and an ambulation score were combined to determine the EDSS steps, ranging from 0 (normal) to 10 (death due to MS). 3-month confirmed disability progression is defined as an increase of score of 1 point in patients with baseline score of 3.0 to 5.0 and 0.5 point increase with baseline score of 5.5 to 6.5 sustained for at least 3 months.
Time Frame: Baseline, every 3 month up to the maximum of approximately 3 years
Population: The Full analysis set (FAS), which comprised all randomized patients with assigned treatments who took at least one dose of study medication, was considered for the analysis. Only participants from the FAS with non-missing covariates were analyzed for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 1096 | 545
Percentage of participants | 26.3 | 31.7
Statistical Analysis 1: Comparison: Siponimod (BAF312) vs Placebo; Test type: Superiority; p = 0.0134, Cox proportional hazards model; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.65 to 0.95]

2. Secondary Outcome: Percentage of Participants With 3-month Confirmed Worsening in T25W of at Least 20% From Baseline
Description: The Timed 25-Foot Walk Test (T25W) measured the time, in seconds, to walk 25 feet (7.62 meters).
  A 3-month confirmed worsening of at least 20% from baseline in the T25W was defined as an increase from baseline sustained for at least 3 months.
  This outcome measure was analyzed using a Cox proportional hazards model.
Time Frame: Baseline, every 3 months up to the maximum of approximately 3 years
Population: Participants from the FAS with non-missing covariates for the model.
Measure: Number; unit: Percentage of participants
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 1087 | 543
Percentage of participants | 39.7 | 41.4
Statistical Analysis 1: Comparison: Siponimod (BAF312) vs Placebo; Test type: Superiority; p = 0.4398, Cox proportional hazards model; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.80 to 1.10]

3. Secondary Outcome: Change From Baseline in T2 Lesion Volume
Description: Magnetic resonance imaging (MRI) scans of the brain were performed every 12 months. MRI evaluation during the Core Part included the total volume of T2 lesions. Each MRI scan was reviewed by a local neurologist and by a central blinded MRI reading center.
  The change from baseline in T2 lesion volume was analyzed using a mixed model for repeated measures (MMRM) with visit as a categorical factor and an unstructured covariance matrix and with adjustment for baseline covariates.
Time Frame: Baseline, Month 12 and Month 24
Population: Participants from the FAS with at least one post-baseline MRI scan and non-missing covariates for the model.
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 995 | 495
mm^3
  Month 12 | 204.9 (67.47) | 818.0 (87.29)
  Month 24 | 162.9 (73.90) | 940.4 (97.20)
  Average over Month 12 and Month 24 | 183.9 (66.33) | 879.2 (85.43)
Statistical Analysis 1: Comparison: Siponimod (BAF312) vs Placebo; Month 12; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -613.1, 95% CI 2-sided [-800.2 to -426.0], Standard Error of Mean 95.39
Statistical Analysis 2: Comparison: Siponimod (BAF312) vs Placebo; Month 24; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -777.5, 95% CI 2-sided [-990.6 to -564.4], Standard Error of Mean 108.62
Statistical Analysis 3: Comparison: Siponimod (BAF312) vs Placebo; Average over Month 12 and Month 24; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -695.3, 95% CI 2-sided [-877.3 to -513.3], Standard Error of Mean 92.79

4. Secondary Outcome: Percentage of Participants With 6-month Confirmed Disability Progression (CDP) Events as Measured by the Expanded Disability Status Scale (EDSS)
Description: The EDSS uses an ordinal scale to assess neurologic impairment in multiple sclerosis (MS) based on a neurological examination. Scores in each of 7 functional systems (Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel & Bladder, and Cerebral) and an ambulation score were combined to determine the EDSS steps, ranging from 0 (normal) to 10 (death due to MS).
  6-month confirmed disability progression is defined as an increase of score of 1 point in patients with baseline score of 3.0 to 5.0 and 0.5 point increase with baseline score of 5.5 to 6.5 sustained for at least 6 months.
  This outcome measure was analyzed using a Cox proportional hazards model.
Time Frame: Baseline, every 3 months up to the maximum of approximately 3 years
Population: Participants from the FAS with non-missing covariates for the model.
Measure: Number; unit: Percentage of participants
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 1096 | 545
Percentage of participants | 19.9 | 25.5
Statistical Analysis 1: Comparison: Siponimod (BAF312) vs Placebo; Test type: Superiority; p = 0.0058, Cox proportional hazards model; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.60 to 0.92]

5. Secondary Outcome: Annualized Relapse Rate (ARR) for Confirmed Relapses
Description: Multiple sclerosis (MS) relapse was defined as appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. Additionally, the abnormality had to be present for at least 24 hours and occur in the absence of fever (<37.5°C) or known infection.
  A confirmed MS relapse was defined as accompanied by a clinically-relevant change in the EDSS, as defined in the study protocol, performed by the Independent EDSS Rater.
  ARR was defined as the average number of confirmed relapses per year. ARR was analyzed using a negative binomial regression model.
Time Frame: Up to maximum approximately 3 years
Population: All participants in the FAS
Measure: Mean (95% Confidence Interval); unit: relapses/year
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 1099 | 546
relapses/year | 0.071 [0.055 to 0.092] | 0.160 [0.123 to 0.207]
Statistical Analysis 1: Comparison: Siponimod (BAF312) vs Placebo; Test type: Superiority; p < 0.0001, Negative binomial regression model; ARR ratio = 0.445, 95% CI 2-sided [0.337 to 0.587]

6. Secondary Outcome: Percentage of Participants With First Relapse Events as Measured by Time to First Confirmed Relapse
Description: Multiple sclerosis (MS) relapse was defined as appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. Additionally, the abnormality had to be present for at least 24 hours and occur in the absence of fever (<37.5°C) or known infection.
  A confirmed MS relapse was defined as accompanied by a clinically-relevant change in the EDSS, as defined in the study protocol, performed by the Independent EDSS Rater.
  Time to first relapse was defined as the time from Day 1 until the start of relapse symptoms. Patients without relapse were censored at the latest known date to be at risk.
  This outcome measure was analyzed using a Cox proportional hazards model.
Time Frame: Up to maximum approximately 3 years
Population: Participants from the FAS with non-missing covariates for the model.
Measure: Number; unit: Percentage of participants
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 1061 | 528
Percentage of participants | 10.7 | 18.9
Statistical Analysis 1: Comparison: Siponimod (BAF312) vs Placebo; Test type: Superiority; p < 0.0001, Cox proportional hazards model; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.41 to 0.70]

7. Secondary Outcome: Percentage of Patients With Relapse (Confirmed Relapse and Any Relapse)
Description: Multiple sclerosis (MS) relapse was defined as appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. Additionally, the abnormality had to be present for at least 24 hours and occur in the absence of fever (<37.5°C) or known infection.
  A confirmed MS relapse was defined as accompanied by a clinically-relevant change in the EDSS, as defined in the study protocol, performed by the Independent EDSS Rater.
Time Frame: Up to maximum approximately 3 years
Population: All participants in the FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 1099 | 546
Percentage of participants
  Any relapse (confirmed or unconfirmed) | 16.7 | 26.0
  Confirmed relapse | 10.3 | 18.7

8. Secondary Outcome: Change From Baseline in MSWS-12 Converted Score
Description: The Multiple Sclerosis Walking Scale (MSWS-12) version 2 is a patient-rated measure of walking consisting of 12 items. Walking limitations were reported by the patients using categories, generating a total transformed score ranging from 0-100. Higher scores reflected greater impairment.
  The change from baseline in MSWS-12 converted score was analyzed using a repeated measures model.
Time Frame: Baseline, Month 12 and Month 24
Population: Participants from the FAS with an available value for the MSWS-12 converted score at baseline and at least one post-baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 1022 | 516
score on a scale
  Month 12 | 1.53 (0.678) | 3.36 (0.908)
  Month 24 | 4.16 (0.848) | 5.38 (1.167)
Statistical Analysis 1: Comparison: Siponimod (BAF312) vs Placebo; Month 12; Test type: Superiority; p = 0.0764, Repeated measures model; Mean Difference (Final Values) = -1.83, 95% CI 2-sided [-3.85 to 0.19], Standard Error of Mean 1.030
Statistical Analysis 2: Comparison: Siponimod (BAF312) vs Placebo; Month 24; Test type: Superiority; p = 0.3671, Repeated measures model; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-3.89 to 1.44], Standard Error of Mean 1.359

9. Secondary Outcome: Number of T1 Gd-enhancing Lesions Per Patient Per Scan
Description: Magnetic resonance imaging (MRI) scans of the brain were performed every 12 months. MRI evaluation during the Core Part included the number of T1 gadolinium (Gd)-enhancing lesions. Each MRI scan was reviewed by a local neurologist and by a central blinded MRI reading center.
  The number of T1 Gd-enhancing lesions per patient per scan was analyzed using a negative binomial regression model.
Time Frame: Baseline, Month 12 and Month 24
Population: Participants from the FAS with at least one post-baseline MRI scan and non-missing values for the covariates included in the model.
Measure: Least Squares Mean (95% Confidence Interval); unit: T1 Gd-enhancing lesions/patient/scan
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 996 | 496
T1 Gd-enhancing lesions/patient/scan
  Month 12 | 0.080 [0.058 to 0.111] | 0.640 [0.488 to 0.839]
  Month 24 | 0.074 [0.040 to 0.138] | 0.418 [0.288 to 0.607]
Statistical Analysis 1: Comparison: Siponimod (BAF312) vs Placebo; Month 12; Test type: Superiority; p < 0.0001, Negative binomial regression model; Rate ratio = 0.126, 95% CI 2-sided [0.083 to 0.191]
Statistical Analysis 2: Comparison: Siponimod (BAF312) vs Placebo; Month 24; Test type: Superiority; p < 0.0001, Negative binomial regression model; Rate ratio = 0.178, 95% CI 2-sided [0.087 to 0.362]

10. Secondary Outcome: Number of New or Enlarging T2 Lesions Per Patient Per Year
Description: Magnetic resonance imaging (MRI) scans of the brain were performed every 12 months. MRI evaluation during the Core Part included the number of new or enlarging T2 lesions. Each MRI scan was reviewed by a local neurologist and by a central blinded MRI reading center.
  The number of new or enlarging T2 lesions compared to previous scan was analyzed using a repeated measures negative binomial regression model.
Time Frame: Baseline, Month 12 and Month 24
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: T2 lesions/patient/year
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 997 | 496
T2 lesions/patient/year
  Month 12 | 1.003 [0.858 to 1.172] | 3.776 [3.148 to 4.528]
  Month 24 | 0.489 [0.371 to 0.644] | 3.437 [2.800 to 4.220]
Statistical Analysis 1: Comparison: Siponimod (BAF312) vs Placebo; Month 12; Test type: Superiority; p < 0.0001, Regression model; Repeated measures negative binomial regression model; Rate ratio = 0.266, 95% CI 2-sided [0.215 to 0.328]
Statistical Analysis 2: Comparison: Siponimod (BAF312) vs Placebo; Month 24; Test type: Superiority; p < 0.0001, Regression model; Repeated measures negative binomial regression model; Rate ratio = 0.142, 95% CI 2-sided [0.103 to 0.196]

11. Secondary Outcome: Percent Brain Volume Change (PBVC) Relative to Baseline
Description: Magnetic resonance imaging (MRI) scans of the brain were performed every 12 months. MRI evaluation during the Core Part included the percentage change in brain volume. Each MRI scan was reviewed by a local neurologist and by a central blinded MRI reading center.
  PBVC relative to baseline was analyzed using a repeated measures model (for normally distributed data) with visit as a categorical factor.
Time Frame: Baseline, Month 12 and Month 24
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: % change from baseline in brain volume
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 894 | 436
% change from baseline in brain volume
  Month 12 | -0.283 (0.0264) | -0.458 (0.0341)
  Month 24 | -0.711 (0.0356) | -0.839 (0.0476)
Statistical Analysis 1: Comparison: Siponimod (BAF312) vs Placebo; Month 12; Test type: Superiority; p < 0.0001, Repeated measures model; Mean Difference (Final Values) = 0.175, 95% CI 2-sided [0.103 to 0.247], Standard Error of Mean 0.0367
Statistical Analysis 2: Comparison: Siponimod (BAF312) vs Placebo; Month 24; Test type: Superiority; p = 0.0196, Repeated measures model; Mean Difference (Final Values) = 0.128, 95% CI 2-sided [0.021 to 0.236], Standard Error of Mean 0.0549

12. Secondary Outcome: Number of Participants With 3-month CDP Events as Measured by EDSS in the Subgroup of SPMS Patients With/Without Superimposed Relapses
Description: The Expanded Disability Status Scale (EDSS) assesses neurologic impairment in multiple sclerosis (MS). EDSS scale ranges from 0 (normal) to 10 (death due to MS). Confirmed disability is defined as an increase of score of 1 point in patients with baseline score of 3.0 to 5.0 and 0.5 point increase with baseline score of 5.5 to 6.5.
  The definition of 3-month confirmed disability progression (CDP) was an increase from baseline in EDSS as defined before sustained for at least 3 months.
  The following secondary progressive multiple sclerosis (SPMS) groups were defined for the analysis of this endpoint:
  * Without superimposed relapses in the 2 years prior to study start (baseline definition)
  * With superimposed relapses in the 2 years prior to study start (baseline definition)
  * Without superimposed relapses during the Core Part of study (post-treatment)
  * With superimposed relapses during the Core Part of study (post-treatment) Data was analyzed using a Cox proportional hazard model
Time Frame: Baseline, every 3 months up to the maximum of approximately 3 years
Population: Participants from the FAS in each subgroup with an available value for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 1099 | 546
Participants
  Without superimposed relapses at baseline: number analyzed (Participants) | 708 | 343
  Without superimposed relapses at baseline | 190 | 101
  With superimposed relapses at baseline: number analyzed (Participants) | 388 | 202
  With superimposed relapses at baseline | 98 | 72
  Without superimposed relapses post-treatment: number analyzed (Participants) | 986 | 444
  Without superimposed relapses post-treatment | 237 | 122
  With superimposed relapses post-treatment: number analyzed (Participants) | 113 | 102
  With superimposed relapses post-treatment | 51 | 51
Statistical Analysis 1: Comparison: Siponimod (BAF312) vs Placebo; Without superimposed relapses at baseline; Test type: Superiority; Cox proportional hazard model; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.68 to 1.11]
Statistical Analysis 2: Comparison: Siponimod (BAF312) vs Placebo; With superimposed relapses at baseline; Test type: Superiority; Cox proportional hazard model; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.49 to 0.91]
Statistical Analysis 3: Comparison: Siponimod (BAF312) vs Placebo; Without superimposed relapses post-treatment; Test type: Superiority; Cox proportional hazard model; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.69 to 1.06]
Statistical Analysis 4: Comparison: Siponimod (BAF312) vs Placebo; With superimposed relapses post-treatment; Test type: Superiority; Cox proportional hazard model; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.53 to 1.19]

13. Secondary Outcome: Number of Participants With 3-month CDP Events as Measured by EDSS in the Subgroup of Rapidly and Not Rapidly Evolving Patients
Description: The Expanded Disability Status Scale (EDSS) assesses neurologic impairment in multiple sclerosis (MS). EDSS scale ranges from 0 (normal) to 10 (death due to MS). Confirmed disability is defined as an increase of score of 1 point in patients with baseline score of 3.0 to 5.0 and 0.5 point increase with baseline score of 5.5 to 6.5.
  The definition of 3-month confirmed disability progression (CDP) was an increase from baseline in EDSS as defined before sustained for at least 3 months.
  Rapidly evolving patients are defined as subjects with 1.5 or greater EDSS change in the 2 years prior to or at study start and disability progression in the 2 years prior to study start was not adjudicated.
  Data was analyzed using a Cox proportional hazard model.
Time Frame: Baseline, every 3 months up to the maximum of approximately 3 years
Population: Participants from the FAS in each subgroup with an available value for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 1099 | 546
Participants
  Rapidly evolving patients: number analyzed (Participants) | 264 | 145
  Rapidly evolving patients | 82 | 60
  Not rapidly evolving patients: number analyzed (Participants) | 835 | 401
  Not rapidly evolving patients | 206 | 113
Statistical Analysis 1: Comparison: Siponimod (BAF312) vs Placebo; Rapidly evolving patients; Test type: Superiority; Cox proportional hazard model; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.46 to 0.91]
Statistical Analysis 2: Comparison: Siponimod (BAF312) vs Placebo; Not rapidly evolving patients; Test type: Superiority; Cox proportional hazard model; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.69 to 1.09]

14. Secondary Outcome: Number of Participants With 3-month CDP Events as Measured by EDSS in the Subgroup of Patients With and Without Moderate/Severe Disease Course
Description: The Expanded Disability Status Scale (EDSS) assesses neurologic impairment in multiple sclerosis (MS). EDSS scale ranges from 0 (normal) to 10 (death due to MS). Confirmed disability is defined as an increase of score of 1 point in patients with baseline score of 3.0 to 5.0 and 0.5 point increase with baseline score of 5.5 to 6.5.
  The definition of 3-month confirmed disability progression (CDP) was an increase from baseline in EDSS as defined before sustained for at least 3 months.
  Moderate or severe course of disease is defined as global Multiple Sclerosis Severity Score (MSSS) of 4 or more at baseline.
  Data was analyzed using a Cox proportional hazard model.
Time Frame: Baseline, every 3 months up to the maximum of approximately 3 years
Population: Participants from the FAS in each subgroup with an available value for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Siponimod (BAF312) | Placebo
Number analyzed (Participants) | 1099 | 546
Participants
  With moderate or severe course of disease: number analyzed (Participants) | 904 | 459
  With moderate or severe course of disease | 232 | 141
  Without moderate or severe course of disease: number analyzed (Participants) | 195 | 87
  Without moderate or severe course of disease | 56 | 32
Statistical Analysis 1: Comparison: Siponimod (BAF312) vs Placebo; With moderate or severe course of disease; Test type: Superiority; Cox proportional hazard model; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.65 to 0.99]
Statistical Analysis 2: Comparison: Siponimod (BAF312) vs Placebo; Without moderate or severe course of disease; Test type: Superiority; Cox proportional hazard model; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.47 to 1.13]

ADVERSE EVENTS:
Time Frame: Core Part: from first dose of double-blind study treatment until end of Core Part (up to approximately 3 years). Core and Extension: from first dose of siponimod until end of study (up to approximately 10 years).
Description: Safety is assessed in the Safety Set, including all patients who received at least one dose of study medication.
  The "All BAF312" group comprises all patients who received at least one dose of siponimod, including those who had 6-month CDP during the Treatment Epoch of the Core Part and received open label siponimod as rescue medication.
Groups:
- Core-BAF312: Participants who were randomized to siponimod (BAF312) during the Core Part
- Core-Placebo: Participants who were randomized to placebo during the Core Part
- All BAF312: All participants who received at least one dose of siponimod (BAF312) during the Core Part and/or the Extension Part
Arm/Group | Core-BAF312 | Core-Placebo | All BAF312
All-Cause Mortality (participants affected / at risk) | 4/1099 | 4/546 | 33/1517
Serious Adverse Events (participants affected / at risk) | 196/1099 | 83/546 | 610/1517
Other Adverse Events (participants affected / at risk) | 778/1099 | 348/546 | 1267/1517
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core-BAF312 (N=1099) | Core-Placebo (N=546) | All BAF312 (N=1517)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 4
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphocytic infiltration (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 4
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 3
Angina pectoris (Cardiac disorders) | 1 | 1 | 3
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 2 | 0 | 2
Bradycardia (Cardiac disorders) | 3 | 0 | 4
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1 | 2
Myocardial infarction (Cardiac disorders) | 0 | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 2
Brugada syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 1
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 1
Malformation venous (Congenital, familial and genetic disorders) | 0 | 0 | 1
Deafness transitory (Ear and labyrinth disorders) | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1
Graves' disease (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Blindness (Eye disorders) | 1 | 0 | 2
Cataract (Eye disorders) | 0 | 1 | 2
Diplopia (Eye disorders) | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 1
Macular hole (Eye disorders) | 0 | 0 | 1
Macular oedema (Eye disorders) | 3 | 0 | 6
Photophobia (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 1
Retinoschisis (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Acquired oesophageal web (Gastrointestinal disorders) | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 3
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 7
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Accidental death (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 2 | 0 | 4
Chills (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 3
Gait disturbance (General disorders) | 1 | 3 | 3
General physical health deterioration (General disorders) | 0 | 0 | 2
Granuloma (General disorders) | 0 | 0 | 1
Hyperpyrexia (General disorders) | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 2
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 11
Sudden cardiac death (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 4
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 5
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 1
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 0 | 1
Abscess soft tissue (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Appendiceal abscess (Infections and infestations) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 3 | 0 | 3
Appendicitis perforated (Infections and infestations) | 0 | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 0 | 2
Bacterial infection (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 3
Burn infection (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 14
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 6
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 3
Central nervous system infection (Infections and infestations) | 0 | 0 | 1
Chorioretinitis (Infections and infestations) | 1 | 0 | 2
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1
Complicated appendicitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 4
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 3
Encephalitis viral (Infections and infestations) | 0 | 0 | 1
Enterovirus infection (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 1 | 7
Gastroenteritis proteus (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Groin abscess (Infections and infestations) | 0 | 0 | 2
Hepatitis E (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 5
Herpes zoster meningitis (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 1 | 6
Labyrinthitis (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 4
Meningitis cryptococcal (Infections and infestations) | 0 | 0 | 2
Nasal abscess (Infections and infestations) | 1 | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 2
Oral viral infection (Infections and infestations) | 1 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 2
Otosalpingitis (Infections and infestations) | 0 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 28
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 4
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 1 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 9
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 15
Septic encephalopathy (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 2 | 0 | 7
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 4
Urinary tract infection (Infections and infestations) | 15 | 7 | 67
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 3
Urosepsis (Infections and infestations) | 5 | 1 | 13
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 8
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bursa injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 5 | 0 | 8
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 3
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 11
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 1 | 13
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2 | 5
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 4
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury corneal (Injury, poisoning and procedural complications) | 1 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 3
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Maisonneuve fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 2
Nerve root injury cervical (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 3
Reactive gastropathy (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Shoulder fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 4 | 0 | 8
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Splenic injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subarachnoid haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 6
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 3
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 10 | 2 | 19
Aspartate aminotransferase increased (Investigations) | 5 | 1 | 9
Blood bilirubin increased (Investigations) | 2 | 0 | 3
Blood glucose increased (Investigations) | 1 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 1
CD8 lymphocytes decreased (Investigations) | 0 | 0 | 1
Columbia suicide severity rating scale abnormal (Investigations) | 2 | 0 | 2
Heart rate decreased (Investigations) | 1 | 0 | 1
Hepatic enzyme abnormal (Investigations) | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 4
Liver function test abnormal (Investigations) | 0 | 1 | 1
Liver function test increased (Investigations) | 0 | 0 | 2
Lung diffusion test decreased (Investigations) | 1 | 0 | 2
Magnetic resonance imaging abnormal (Investigations) | 0 | 0 | 1
Pulmonary function test decreased (Investigations) | 1 | 0 | 2
Troponin increased (Investigations) | 0 | 0 | 1
Walking distance test abnormal (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 4
Haemochromatosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemic crisis (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Shock hypoglycaemic (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Ligament disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 9
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 7 | 68
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 18
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 7
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 6
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 4
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 3
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 8
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 10
Squamous cell carcinoma of the vagina (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 6
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Allodynia (Nervous system disorders) | 0 | 1 | 0
Amnestic disorder (Nervous system disorders) | 0 | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0 | 2
Ataxia (Nervous system disorders) | 1 | 0 | 2
Autoimmune demyelinating disease (Nervous system disorders) | 0 | 0 | 1
Brain injury (Nervous system disorders) | 1 | 0 | 1
Brain stem infarction (Nervous system disorders) | 1 | 0 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 2
Cerebral infarction (Nervous system disorders) | 0 | 0 | 3
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 7
Clonic convulsion (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 3
Epilepsy (Nervous system disorders) | 5 | 0 | 22
Facial paresis (Nervous system disorders) | 0 | 0 | 1
Febrile infection-related epilepsy syndrome (Nervous system disorders) | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 3
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0
Head titubation (Nervous system disorders) | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 3 | 0 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Hypokinesia (Nervous system disorders) | 0 | 0 | 1
Intention tremor (Nervous system disorders) | 1 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 4
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1
Lacunar stroke (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Meralgia paraesthetica (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 2
Migraine with aura (Nervous system disorders) | 0 | 0 | 1
Motor dysfunction (Nervous system disorders) | 0 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 2 | 0 | 17
Multiple sclerosis pseudo relapse (Nervous system disorders) | 0 | 0 | 3
Multiple sclerosis relapse (Nervous system disorders) | 2 | 7 | 7
Muscle spasticity (Nervous system disorders) | 2 | 1 | 9
Optic neuritis (Nervous system disorders) | 0 | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 3 | 2
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 2 | 0 | 6
Polyneuropathy (Nervous system disorders) | 1 | 0 | 2
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1
Postictal paralysis (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 2
Progressive multiple sclerosis (Nervous system disorders) | 0 | 0 | 1
Pseudobulbar palsy (Nervous system disorders) | 0 | 0 | 1
Putamen haemorrhage (Nervous system disorders) | 0 | 1 | 0
Quadriparesis (Nervous system disorders) | 0 | 0 | 2
Quadriplegia (Nervous system disorders) | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0 | 1
Secondary progressive multiple sclerosis (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 4 | 0 | 7
Status epilepticus (Nervous system disorders) | 0 | 0 | 4
Status migrainosus (Nervous system disorders) | 1 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Subdural hygroma (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 4 | 1 | 6
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 6
Tremor (Nervous system disorders) | 0 | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 3 | 0 | 12
Uhthoff's phenomenon (Nervous system disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 2
Device breakage (Product Issues) | 0 | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 2
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 1 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 4
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 3 | 2 | 3
Depression suicidal (Psychiatric disorders) | 1 | 0 | 1
Depressive symptom (Psychiatric disorders) | 1 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 3
Drug abuse (Psychiatric disorders) | 0 | 0 | 1
Euphoric mood (Psychiatric disorders) | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Major depression (Psychiatric disorders) | 0 | 0 | 1
Mania (Psychiatric disorders) | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 1
Mixed anxiety and depressive disorder (Psychiatric disorders) | 2 | 0 | 2
Panic attack (Psychiatric disorders) | 1 | 1 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 2
Suicidal behaviour (Psychiatric disorders) | 3 | 0 | 4
Suicidal ideation (Psychiatric disorders) | 3 | 1 | 8
Suicide attempt (Psychiatric disorders) | 4 | 3 | 8
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 5
Bladder dysfunction (Renal and urinary disorders) | 2 | 0 | 3
Bladder hypertrophy (Renal and urinary disorders) | 0 | 0 | 2
Bladder leukoplakia (Renal and urinary disorders) | 0 | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 2
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 2
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 1 | 2
Nephritis (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 4
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 1 | 0 | 2
Obstructive nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1
Single functional kidney (Renal and urinary disorders) | 1 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 3
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 1
Urge incontinence (Renal and urinary disorders) | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 3
Urinary retention (Renal and urinary disorders) | 3 | 2 | 9
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 2
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 2
Heavy menstrual bleeding (Reproductive system and breast disorders) | 2 | 0 | 3
Intermenstrual bleeding (Reproductive system and breast disorders) | 2 | 1 | 2
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian disorder (Reproductive system and breast disorders) | 1 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1
Testicular atrophy (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 8
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5
Respiratory paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Actinic elastosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 4
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Immobile (Social circumstances) | 1 | 0 | 1
Walking disability (Social circumstances) | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 5
Essential hypertension (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 2
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Internal haemorrhage (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core-BAF312 (N=1099) | Core-Placebo (N=546) | All BAF312 (N=1517)
Lymphopenia (Blood and lymphatic system disorders) | 9 | 0 | 137
Constipation (Gastrointestinal disorders) | 39 | 21 | 103
Diarrhoea (Gastrointestinal disorders) | 69 | 22 | 119
Nausea (Gastrointestinal disorders) | 73 | 19 | 119
Fatigue (General disorders) | 100 | 51 | 171
Oedema peripheral (General disorders) | 50 | 13 | 107
Bronchitis (Infections and infestations) | 36 | 16 | 94
COVID-19 (Infections and infestations) | 0 | 0 | 189
Cystitis (Infections and infestations) | 28 | 13 | 79
Herpes zoster (Infections and infestations) | 24 | 4 | 92
Influenza (Infections and infestations) | 72 | 40 | 152
Nasopharyngitis (Infections and infestations) | 149 | 79 | 325
Upper respiratory tract infection (Infections and infestations) | 89 | 41 | 165
Urinary tract infection (Infections and infestations) | 128 | 75 | 369
Contusion (Injury, poisoning and procedural complications) | 34 | 15 | 96
Fall (Injury, poisoning and procedural complications) | 126 | 59 | 295
Alanine aminotransferase increased (Investigations) | 58 | 8 | 108
Gamma-glutamyltransferase increased (Investigations) | 43 | 6 | 120
Lymphocyte count decreased (Investigations) | 4 | 0 | 84
Hypercholesterolaemia (Metabolism and nutrition disorders) | 28 | 11 | 99
Arthralgia (Musculoskeletal and connective tissue disorders) | 69 | 42 | 184
Back pain (Musculoskeletal and connective tissue disorders) | 65 | 43 | 186
Pain in extremity (Musculoskeletal and connective tissue disorders) | 60 | 21 | 113
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 45 | 15 | 130
Dizziness (Nervous system disorders) | 74 | 26 | 145
Headache (Nervous system disorders) | 158 | 71 | 249
Muscle spasticity (Nervous system disorders) | 41 | 23 | 89
Depression (Psychiatric disorders) | 43 | 28 | 134
Insomnia (Psychiatric disorders) | 37 | 19 | 84
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 18 | 90
Actinic keratosis (Skin and subcutaneous tissue disorders) | 15 | 6 | 80
Hypertension (Vascular disorders) | 114 | 41 | 294

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.